CLINICAL TRIAL: NCT03065816
Title: A Randomized, Open-label, 2-Treatment Crossover Study to Compare by Scintigraphy, the Antireflux Activity of the To-be-Registered Product (250 mg Sodium Alginate/187.5 mg Calcium Carbonate/106.5 mg Sodium Hydrogen Carbonate) Chewable Tablets Versus the Registered Gaviscon Double Action Tablets, in Healthy Adult Subjects
Brief Title: Scintigraphy Study to Compare the Antireflux Activity of the Z0063 Versus Gaviscon Double Action Tablets, in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: PDY14363; 2015-000764-34 (EudraCT Number); U1111-1182-1864 (Other: UTN)
Record Dates: First submitted 2017-02-23; First posted 2017-02-28 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Gastroesophageal Reflux Disease
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — alginate, aluminium hydroxide, magnesium trisilicate, sodium bicarbonate drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence 1 (Z0063 to Gaviscon) (Experimental): The subjects will be given Z0063 single dose and then will crossover to Gaviscon single dose
  Interventions: Drug: Z0063; Drug: Gaviscon
- Sequence 2 (Gaviscon to Z0063) (Experimental): The subjects will be given Gaviscon single dose and then will crossover to Z0063 single dose
  Interventions: Drug: Z0063; Drug: Gaviscon

INTERVENTIONS:
Drug: Z0063 — Pharmaceutical form: chewable tablets Route of administration: oral
Drug: Gaviscon — Pharmaceutical form: chewable tablets Route of administration: oral

SUMMARY:
Primary Objective:

Pharmacodynamics: assessment and comparison by gamma scintigraphy of the gastric retention of alginate rafts (raft performance) of Z0063 to the effect of Gaviscon Double Action Tablets, in healthy adult subjects.

Secondary Objective:

Safety: assessment of the clinical safety of Z0063 versus Gaviscon Double Action tablets, in healthy adult subjects.

DETAILED DESCRIPTION:
The total study duration per subject is 37 days including a screening period up to 21 days, a wash-out period of 4-7 days and a follow-up of 4-7 days.

ELIGIBILITY:
Inclusion criteria :

* Male or female subjects, between 18 and 55 years of age, inclusive.
* Body weight between 50.0 and 100.0 kg, inclusive, if male, and between 40.0 and 90.0 kg, inclusive, if female, body mass index between 18.0 and 28.0 kg/m^2, inclusive.
* Certified as healthy by a comprehensive clinical assessment.
* Normal vital signs, electrocardiogram (ECG) and laboratory parameters.
* Subject has to be willing to eat the standard radiolabelled meal (eggs on toasts and orange juice).

Exclusion criteria:

* Any history or presence of clinically relevant abnormalities at screening which could interfere with the objectives of the study or the safety of the subject's participation.
* Blood donation of more than 450 mL within 3 months before inclusion.
* History or presence of drug or alcohol abuse.
* Smoking more than 5 cigarettes or equivalent per day, unable to stop smoking during the study.
* If female, pregnancy (defined as positive beta-human chorionic gonadotropin [β-HCG] blood test), breast-feeding.
* Any medication (including St John's Wort) within 14 days before inclusion with the exception of hormonal contraception or menopausal hormone replacement therapy.
* Any subject in the exclusion period of a previous study: participation in a new chemical entity clinical study within the previous 3 months or a marketed drug clinical study within the previous 30 days.
* Any subject who cannot be contacted in case of emergency.
* Positive result on any of the following tests: hepatitis B surface (HBs Ag) antigen, anti-hepatitis C virus (anti-HCV) antibodies, anti-human immunodeficiency virus 1 and 2 antibodies (anti-HIV1 and anti HIV2 Ab).
* Positive result on urine drug screen.
* Positive alcohol test.
* Known hypersensitive to alginates, products or formulation excipients and/or to any component of the standardized meal.
* Any subject with difficulty in chewing and/or swallowing.
* Participation in a study in which radioisotopes were administered or in which subject was exposed to any radiation other than normal background radiation within the 12 months before the screening visit.
* Any intake of aluminum and magnesium containing antacids or other alginate-containing medicinal products within 14 days before inclusion.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2017-02-09 (Actual); Primary Completion 2017-05-02 (Actual); Study Completion 2017-05-02 (Actual)

PRIMARY OUTCOMES:
Pharmacodynamics: area under curve (AUC) of investigational medicinal product (IMP) percentage retention in the whole stomach | 4 hours after IMP administration

SECONDARY OUTCOMES:
Pharmacodynamics: AUC of meal percentage retention in the whole stomach | 4 hours after IMP administration

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational site 826001, Merthyr Tydfil, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org